CLINICAL TRIAL: NCT02998840
Title: A Prospective, Vehicle Controlled, Double Blinded, Multicenter, Randomized, Phase II Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects With Elevated Blood Pressure
Brief Title: A Prospective Study of B244 Delivered as a Topical Spray to Determine Safety and Efficacy in Subjects With Elevated Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AOBiome LLC (Industry)
Collaborators: Veristat, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVB244-003
Record Dates: First submitted 2016-11-22; First posted 2016-12-21 (Estimated); Results first posted 2022-08-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Prehypertension; Hypertension, Stage I
Keywords: elevated blood pressure
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- B244 4 pumps applied to the face (Active Comparator): 4 pumps total of spray to saturate the entire face. Applications should occur in the morning and at night for 4 weeks.
  Interventions: Biological: B244
- B 244 8 Pumps applied to face and torso (Active Comparator): 8 pumps total - 4 pumps of spray to saturate the entire face and 4 pumps to the torso Applications should occur in the morning and at night for 4 weeks.
  Interventions: Biological: B244
- Vehicle 4 pumps applied to the face (Sham Comparator): 4 pumps total of spray to saturate the entire face. Applications should occur in the morning and at night for 4 weeks.
  Interventions: Biological: Vehicle
- Vehicle 8 pumps applied to face and torso (Sham Comparator): 8 pumps total - 4 pumps of spray to saturate the entire face and 4 pumps to the torso Applications should occur in the morning and at night for 4 weeks.
  Interventions: Biological: Vehicle

INTERVENTIONS:
Biological: B244 — odorless suspension
  Arms: B 244 8 Pumps applied to face and torso; B244 4 pumps applied to the face
Biological: Vehicle — odorless suspension
  Arms: Vehicle 4 pumps applied to the face; Vehicle 8 pumps applied to face and torso

SUMMARY:
The purpose of this study is to evaluate and compare the efficacy of B244 in treating patients with hypertension.

DETAILED DESCRIPTION:
This is a Prospective, Vehicle Controlled, Double Blinded, Multicenter, Randomized Phase II trial, comparing the effect of twice daily B244 application for 4 weeks vs vehicle application on BP and inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age
* In good general health as determined by a thorough medical history and physical examination, and vital signs
* Clinical diagnosis of elevated Blood Pressure defined as:

  * Having systolic prehypertension measurements having systolic BP (mmHg) of 120-139 and Diastolic BP (mmHg) of 90
  * OR
  * Having systolic Stage 1 hypertension measurements having systolic BP (mmHg) of 140-159 and Diastolic BP (mmHg) of 100
* Hypertension treatment naïve patients, defined as those patients who have never been treated with antihypertensive medications or have been off any hypertensive treatment for a period of 12 weeks or longer.
* Willing to refrain from using any antihypertensive treatments, other than the investigational product, including herbal supplements, systemic use of steroids, chronic use of NSAIDS, any antihypertensive agents, such as beta-blockers, diuretics, ACE inhibitors, CA channel blockers, Alpha blockers, Central Acting agents and vasodilators.
* Ability to comprehend and comply with procedures
* Agree to commit to participate in the current protocol
* Provide written informed consent prior to any study procedure being performed (all subjects should be able to understand the informed consent form and any other documents that subjects are required to read)

Exclusion Criteria:

* Pregnant and/or lactating women
* Patients on treatment for Benign Prostatic Hyperplasia (BPH)
* Clinically significant history of cardiovascular disease (i. e. PCI, CABG MI (if event occurred 12 months), atrial fibrillation, frequent PAC, cardiac rhythm disorder, syncope, valve repair/replacement, heart transplantation, PTA, peripheral bypass surgery, endarterectomy, unstable angina, TIA, stroke and NYHF category II, II and IV heart failure.
* Patients with renal failure, significant kidney or renal disease defined as having creatinine level of mg/dL
* Presence of any condition (medical, psychological, social, or geographical), actual or anticipated, that the Investigator feels would restrict or limit the patient's successful participation for the duration of the study
* History of migraines and/or anxiety, where patient is unable to refrain from the use of beta blockers
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* The participant has been previously randomized in this study
* Subjects with clinical diagnosis of Type I Diabetes
* Subjects with arm circumference of 42 cm
* Any condition that would prevent the subject from participating in the trial in the opinion of the evaluation physician
* The participant has received an investigational product within 30 days prior to randomization
* Prior use of any product containing B244 or Nitrosomonas eutropha
* Unable to lie flat or sit for 15 minutes
* Concurrent participation in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Weiss, MD, Study Director — Chief Medical Officer
Locations (10):
- United States (10):
  - Central Research Associates, Birmingham, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Orange County Research Center, Tustin, California
  - Clinical Research Consulting, Milford, Connecticut
  - AGA Clinical Trials, Hialeah, Florida
  - ICCT Research International, Chicago, Illinois
  - MedPharmics, Metairie, Louisiana
  - Alternative Primary Care (Einstein Clinical Research), Silver Spring, Maryland
  - CHEAR Center, The Bronx, New York
  - Research Trials WorldWide, Humble, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B244 4 Pumps Applied to the Face: 4 pumps total of spray to saturate the entire face. Applications should occur in the morning and at night for 4 weeks.
  B244: odorless suspension, 8x10E9 cells/mL
- B 244 8 Pumps Applied to Face and Torso: 8 pumps total - 4 pumps of spray to saturate the entire face and 4 pumps to the torso Applications should occur in the morning and at night for 4 weeks.
  B244: odorless suspension, 8x10E9 cells/mL
Period: Overall Study
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Vehicle 4 Pumps Applied to the Face | Vehicle 8 Pumps Applied to Face and Torso
Started | 33 | 33 | 33 | 33
Completed | 29 | 30 | 31 | 28
Not Completed | 4 | 3 | 2 | 5
Not completed — Lost to Follow-up | 1 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1
Not completed — Unplanned travel, family emergency, sponsor request, work schedule | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population (ITT): All randomized subjects, analyzed according to treatment assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Vehicle 4 Pumps Applied to the Face | Vehicle 8 Pumps Applied to Face and Torso | Total
Number analyzed (Participants) | 33 | 33 | 33 | 33 | 132
Age, Customized [Count of Participants; unit: Participants]
  <60 years | 25 | 23 | 25 | 27 | 100
  ≥60 years | 8 | 10 | 8 | 6 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 13 | 17 | 62
  Male | 18 | 16 | 20 | 16 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 11 | 12 | 38
  Not Hispanic or Latino | 24 | 27 | 22 | 21 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 13 | 6 | 9 | 36
  White | 23 | 19 | 26 | 22 | 90
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 89.32 (21.084) | 89.04 (21.654) | 86.56 (12.251) | 88.59 (18.871) | 88.38 (18.654)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.139 (6.2438) | 30.427 (5.9047) | 29.306 (4.3707) | 30.304 (6.3886) | 30.044 (5.7332)
BMI Category [Count of Participants; unit: Participants]
  <30 kg/m^2 | 19 | 16 | 20 | 22 | 77
  ≥30 kg/m^2 | 14 | 17 | 13 | 11 | 55
Smoking History [Count of Participants; unit: Participants]
  Never | 19 | 22 | 22 | 19 | 82
  Former | 6 | 7 | 6 | 3 | 22
  Current | 8 | 4 | 5 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Safety and tolerability endpoints will consist of all treatment related adverse events reporting during the study duration.
Time Frame: Baseline-6 weeks
Population: Safety Population: All subjects who received at least 1 dose of study medication. Subjects were to be analyzed according to the study drug received.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps): 4 or 8 pumps total of spray to saturate the entire face (and torso for 8 pumps). Applications should occur in the morning and at night for 4 weeks.
  Vehicle: odorless suspension
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps)
Number analyzed (Participants) | 33 | 33 | 66
Participants
  At Least 1 Treatment Related TEAE | 1 | 1 | 4
  At Least 1 Treatment Related Serious TEAE | 0 | 0 | 0

2. Primary Outcome: Difference in Mean in Clinic Systolic BP Between the Active and Vehicle Groups
Description: Clinical systolic blood pressure (BP) readings were obtained at every visit using a calibrated electronic sphygmomanometer. Three measurements were taken at each visit. The average of the second and third readings was documented. Data was analyzed using mixed-effects model repeated measures (MMRM). Difference was calculated as the change from Baseline to Day 28.
Time Frame: Baseline-Week 4
Population: Subjects from the Intent to Treat (ITT) population (all randomized subjects, analyzed according to treatment assigned) that remained in the study at Week 4.
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps)
Number analyzed (Participants) | 29 | 30 | 61
mmHg | -2.61 (1.828) | -0.66 (1.834) | -2.93 (1.296)

3. Secondary Outcome: Difference in Mean in Clinic Diastolic BP Between the Active and Vehicle Group
Description: Clinical diastolic blood pressure (BP) readings were obtained at every visit using a calibrated electronic sphygmomanometer. Three measurements were taken at each visit. The average of the second and third readings was documented. Data was analyzed using mixed-effects model repeated measures (MMRM). Difference was calculated as the change from Baseline to Day 28.
Time Frame: Baseline-Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps)
Number analyzed (Participants) | 29 | 30 | 61
mmHg | -1.65 (1.377) | -2.25 (1.358) | -1.31 (0.975)

4. Secondary Outcome: Difference in Mean Ambulatory Systolic and Diastolic Daytime Blood Pressure
Description: An ambulatory blood pressure measurement (ABPM) device was placed on a subject's arm during the clinic visit to record 24-hour blood pressure and heart rate measurements.
Time Frame: Baseline-Week 4
Population: Ambulatory Blood Pressure Monitoring Population (ABPP): Subjects in the Safety Population who had valid baseline and Day 28 ambulatory BP monitoring (ABPM) measurements. Subjects who repeated the ABPM were to be included in the population if the repeated assessment met the device monitor's criteria for "passing".
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps)
Number analyzed (Participants) | 29 | 29 | 58
mmHg
  Systolic Blood Pressure | -3.06 (9.388) | -0.21 (12.250) | -0.53 (7.619)
  Diastolic Blood Pressure | -2.17 (5.327) | -0.82 (7.325) | -0.98 (5.911)

5. Other Pre Specified Outcome: Difference in Inflammatory Biomarkers Between Active and Vehicle Groups
Description: To evaluate if B244 administration on the skin twice daily will affect the levels of immune biomarkers.
Time Frame: Baseline-Week 4
Population: Intent to Treat Population (ITT): All randomized subjects, analyzed according to treatment assigned.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps)
Number analyzed (Participants) | 33 | 33 | 66
units on a scale | NA (NA) — NA Explanation: Data not collected/completed for exploratory endpoint. | NA (NA) — NA Explanation: Data not collected/completed for exploratory endpoint. | NA (NA) — NA Explanation: Data not collected/completed for exploratory endpoint.

6. Other Pre Specified Outcome: Microbial Content
Description: Evaluate if B244 administration on skin twice daily will affect the microbial content on collected skin swab samples.
Time Frame: Baseline, Day 28, Day 42
Population: Data was not collected for this exploratory endpoint.
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps)
Number analyzed (Participants) | 0 | 0 | 0

7. Other Pre Specified Outcome: Microbial Composition
Description: Evaluate if B244 administration on skin twice daily will affect the microbial composition on collected skin samples.
Time Frame: Baseline, Day 28, Day 42
Population: Data was not collected for this exploratory endpoint.
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline-Week 6
Description: Participants will report adverse events immediately to the Investigator and study personnel. A safety assessment will be performed at each visit. All adverse events (AEs) recorded during the study through the date of randomization through 28 days after the last dose of study drug will be analyzed.
Arm/Group | B244 4 Pumps Applied to the Face | B 244 8 Pumps Applied to Face and Torso | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/33 | 0/66
Other Adverse Events (participants affected / at risk) | 4/33 | 6/33 | 11/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 4 Pumps Applied to the Face (N=33) | B 244 8 Pumps Applied to Face and Torso (N=33) | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps) (N=66)
Exacerbation of depression (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B244 4 Pumps Applied to the Face (N=33) | B 244 8 Pumps Applied to Face and Torso (N=33) | Pooled Vehicle 4 or 8 Pumps Applied to the Face (and Torso for 8 Pumps) (N=66)
Dizziness (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 1
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 1
Weight increased (Investigations) | 1 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall have 45 days to review the papers. Sponsor shall have the right to require Institution/Principal Investigator, as applicable, to remove specifically identified confidential information and/or delay the proposed publication or presentation for an additional one hundred twenty (120) days to enable Sponsor to seek patent protections.

DOCUMENTS (2):
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT02998840/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT02998840/SAP_001.pdf